CLINICAL TRIAL: NCT00503334
Title: Efficacy and Tolerability of a Preoperative Oral Nutritional Supplement (preOP Booster) Versus Placebo in Visceral Surgery
Brief Title: Preoperative Oral Nutritional Supplement (preOP Booster) in Visceral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Dr. Steffen Benzing, Fresenius Kabi Deutschland GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: N-POB-03-IT
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-11

CONDITIONS: Enteral Nutrition (Food for Special Medical Purposes)
MeSH Terms: interventions — Dietary Supplements; Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- preOP booster (Experimental)
  Interventions: Dietary Supplement: preOP booster (oral nutritional supplement, food for special medical purposes)
- preOP booster placebo (Placebo Comparator)
  Interventions: Dietary Supplement: preOP booster (oral nutritional supplement, food for special medical purposes)

INTERVENTIONS:
Dietary Supplement: preOP booster (oral nutritional supplement, food for special medical purposes) — 3x1 dosage pre-operatively

SUMMARY:
The purpose of this pilot study is to investigate the effect of an oral nutritional supplement (preOP booster) versus placebo regarding metabolic criteria in patients undergoing elective pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective pancreaticoduodenectomy

Exclusion Criteria:

* Concomitant chemotherapy
* Severe malnutrition (SGA score C)
* Conditions affecting gastric emptying

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
laboratory measurements: total endogenous antioxidant capacity, free radicals, CRP; | up to 30 days after surgery

SECONDARY OUTCOMES:
postoperative complications, pre- and postoperative discomfort (well-being), muscle strength at 7 days post-op, length of stay (hospital / ICU), ambulation time, gastro intestinal tolerance | up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marco Braga, Prof MD, Principal Investigator — Università Salute-Vita San Raffaele, Milan, Italy
Locations (1):
- Università Salute-Vita San Raffaele,, Milan, Italy